CLINICAL TRIAL: NCT03831841
Title: Physical Fitness Body Composition and Frailty in Elderly People Above 65 Years. Mediation of Vitamin D and Exercise Program Effects. EXERNET Elder 3.0
Brief Title: Physical Fitness, Body Composition and Frailty in Elderly People.Exercise Program Effecsts. EXERNET Elder 3.0
Acronym: EXERNETElder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, German Vicente-Rodríguez, Senior lecturer, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXERNET Elder 3.0
Record Dates: First submitted 2018-12-02; First posted 2019-02-06 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Frail Elderly Syndrome; Sarcopenia; Physical Activity
Keywords: elderly; multicomponent exercise; body composition; vitamin D; fitness
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multicomponent exercise programe involving all physical fitness paramenters and consisting on sesions of 1 hour, 3 days a week.
  Interventions: Behavioral: Multicomponent exercise programe
- Control (No Intervention): Control group with no intervention programe

INTERVENTIONS:
Behavioral: Multicomponent exercise programe — An intervention consisting of training by a multicomponent program 3 times a week, working on aerobic capacity, flexibility, balance and strength.
  Arms: Intervention

SUMMARY:
One of the major changes occurring in developed societies is a significant ageing of the population. Nowadays, because of an enhanced life expectancy, 17% of the Spanish population is composed of people over 65 and the number is expected to rise to 33% in 2050. Aging is characterized by a gradual lifelong accumulation of molecular and cellular damage that results in a progressive and generalized impairment in several bodily functions, an increased vulnerability to environmental challenges and a growing risk of disease and risk of death. These facts led to an increase on the prevalence of diseases such as osteoporosis diabetes, sarcopenia, obesity or frailty. However, lifestyles such as physical activity could attenuated aging process, maintaining the autonomy of elders, and it has been demonstrated that even implying guided exercise programs could reverse this condition of frailty and dependence.

In this way, the main aims of this research project are to analyze the effect of a multicomponent exercise program in frailty and pre-frailty people above 65 years and without cognitive impairment. Thus, it is going to be evaluated at the beginning and the end of the study; body composition, physical fitness, blood parameters including vitamin D and other health related parameters included in a questionnaire. Secondly, to study the perdurability of training-related gains over time.

DETAILED DESCRIPTION:
The training will consist in a multicomponent exercise program, 3 days a week (Monday, Wednesday and Friday). It will take place during morning in groups of 10-14 and trainers will be qualified. Alll the exercise will be adapted for different levels of frailty and for their functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Above 65 years
* frailty of pre-frailty by SPPB.

Exclusion Criteria:

* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Change in SPPB | Change from Baseline at 3 months, 6 months and 12 months
  Short Physical Performance Battery by Romberg (SPPB): consist of walking 4m, a balance test with three levels (tandem, semi-tandem and stand up on one foot) and sit up and reach 5 times as fast as possible. Each test could point from 0 to 4, reaching a maximum of 12 months in the battery. Puntuation correspond to; 0-4 points the person is not valid, from 4 to 6 frails and form 7-9 pre-frailt
Change in Senior fitness test physical performance battery | Change from Baseline at 3 months, 6 months and 12 months
  A fitness test battery in order to measured physical performance of elderly, it includes: flamingos test (for balance), 30m of walking speed, 30 seconds of sit and reach (strength of lower extremities), 30sconds of arm curl, 6 minutes test (aerobic capacity), sit-up and go test (agility), flexibility of upper and lower extremities. Results are registered without puntuation.
Change of 25-OH Vitamin D concentrations | Change from Baseline at 3 months, 6 months and 12 months
  25-OH Vitamin D concentration in blood test

SECONDARY OUTCOMES:
Changes on Fried Scale | Change from Baseline at 3 months, 6 months and 12 months
  Fried frailty phenotype criteria; measured by 3 questiones (exhaustion, walking more than 2 or 2,5 jours a week (for men or women)a and to have lose weigth (4,5kg) in the last year), Handgrip and 4,5 meters walking. Those who point 2 or 3 are prefrail and 3 or more frail.
Changes on Leucocites | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (%)
Changes on Linfocites | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (%)
Changes on hemoglobine | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (%)
Changes on platelets | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (10^3/uL)
Changes on calcium | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on Cholesterol | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on HDL-Cholesterol | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on LDL-Cholesterol | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on Trigicerids | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on uric acid | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on urea | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on creatine | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on creatine kinasa | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (U/dL)
Changes on glucose | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on lactate deydrogenase | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (UI/dL)
Changes on potasium | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mEq/dL)
Changes on magnesium | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on transferrine | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on albumin | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (g/dL)
Changes on protein c reative | Change from Baseline at 3 months, 6 months and 12 months
  Measured by blood test (mg/dL)
Changes on Bone mass and structure by perifereal quantitative computed tomography | Change from Baseline at 3 months, 6 months and 12 months
  Mass and structure of tibia (at 4, 38, 66 % slides) and radius (4, 66 % slides) by pQCT
Changes on hip perimeter | Change from Baseline at 3 months, 6 months and 12 months
  Hip perimeter measured following ISAK protocol. Centimeters
Change on wrist perimeter | Change from Baseline at 3 months, 6 months and 12 months
  Wrist perimeter following ISAK protocol. Centimeters
Change on calf perimeter | Change from Baseline at 3 months, 6 months and 12 months
  Calf perimeter following ISAK protocol. Centimeters
Changes on arm relaxed perimeter | Change from Baseline at 3 months, 6 months and 12 months
  Calf perimeter following ISAK protocol. Centimeters
Changes on weight | Change from Baseline at 3 months, 6 months and 12 months
  Change on kilograms by bioimpedance measurement (TANITA)
Changes on body fat | Change from Baseline at 3 months, 6 months and 12 months
  Change on kilograms by bioimpedance measurement (TANITA)
Changes on efat percentage | Change from Baseline at 3 months, 6 months and 12 months
  Change on % by bioimpedance measurement (TANITA)
Changes on height | Change from Baseline at 3 months, 6 months and 12 months
  Change on height (cm)
Changes on Unkle-Brachial Index | Change from Baseline at 3 months, 6 months and 12 months
  Vascular measure to observed blood circultaion. With a Doppler, sistolic blood pressure measured in brachial arteries (humerus) and unkle arteries are measured. Then, ratio is calculated dividing both results.
Changes on FRAIL Scale | Change from Baseline at 3 months, 6 months and 12 months
  5 questions scale asking about; lose a 5% of own weigth in the last year, to have more than 5 diseases between cancer, diabetes, chloresterol, asthma, EPOC, IAM, cardiac insuficiency, arthritis, ACVA, ERC, angina, hipertension), exhaustion in the last 4 weeks ,ability to walk 10 steps without help, ability to walk more than 100 meters without help. Confirm 3 or more items means to be frail.
Changes on Clinical frailty scale | Change from Baseline at 3 months, 6 months and 12 months
  A descriptive scale about disability and funcional assessments. Is a practical and efficient tool for assessing frailty. It is compound of 9 options describing stages functionality depending on how much help they need for daily activities (1- very fit, 2- well, 3- managing well, 4- vulnerable, 5- mildly frail, 6- moderately frail, 7- severely frail, 8-very severely frail, 9- terminally ill). One option have to be selected.
Changes on Sociotype Questionnaire for geriatric population | Change from Baseline at 3 months, 6 months and 12 months
  Questionnaire about how people stablish their relationships between three social dimensions (family, friendship, and acquaintance). The questionnaire consisted of 12 questions which point from 0 to 5, having the high punctuation a positive meaning. Final mark is obtained from de sum up pf every point of each question.
Changes on Physical Activity Questionnnaire for the Elder (PASE) | Change from Baseline at 3 months, 6 months and 12 months
  Physical activity questionnaire to assesed daily light, moderate and vigorous physical activities. Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in persons age 65 years and older. The PASE score combines information on leisure, household and occupational activity. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. A total of 10 questions using frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity. Contribution of each questionnaire item to the overall PASE score is determined by the product of the sample mean and activity weight
Changes on Insomnia Severity Index Score | Change from Baseline at 3 months, 6 months and 12 months
  The Insomnia Severity Index (ISI) is a short instrument developed to assess insomnia severity Seven questions asking severity of difficulties to falling asleep, staying asleep, waking up too much early, how unsatisfied the person is with his sleep, how affect daily if there is a problem of sleep life. Severity must be pointed from 0 to 4 and the sum up of all question is calculated for the final mark. 0-7 lack of insomnia, 8-14 subclinical insomnia, 15-21 clinical insomnia (mild), 22-28 clinical insomnia (grave)
Changes on Incontinence Urinary Questionnaire | Change from Baseline at 3 months, 6 months and 12 months
  Questionnaire about urinary incontinence, how it affects they daily life pointing from 1 to 10 (being 10 too much worry) and when it happens. This question does not point, they are only registered.
Changes on EUROQOL (EQ-5D) | Change from Baseline at 3 months, 6 months and 12 months
  EQ-5D is a standardised measure of health status developed in order to provide a simple, generic measure of health for clinical and economic appraisal. It descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. The second part of the questionnire records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents. It should be noted that the numerals 1-3 have no arithmetic properties and should not be used as a cardinal score.
Changes on Use of hospital Resources | Change from Baseline, 6 months and 12 months
  Descriptive measure. Registration through the hospital internet private platform of; medication of the patient, number of medical appointments, number of specialised complementary tests, and other medical resourse that could be used by the patient related to healthcare system.
Change Lawton and Brody Index | Change from Baseline at 3 months, 6 months and 12 months
  Questionnaire about instrumental activities of daily life; Ability to Use Telephone Shopping, Laundry, Mode of Transportation, Food Preparation, Responsibility for Own Medications, Housekeeping and Ability to Handle Finances. Each part has 4 options to tick in order of independent to more dependent. Highest mark is 8 and correspond to a summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Changes on Barthel Index | Change from Baseline at 3 months, 6 months and 12 months.
  Questionnaire about authonomy and dependence in; Feeding, Bathing , Grooming , Dressing , Bowel control , Bladder control , Toilet use , Transfers (bed to chair and back) (, Mobility on level surfaces , Stairs. Puntuation correspond to Independent +10points, Needs help+5points, Unable 0 points). Maximal puntuation is 100.which means independence.
Change on Risk of falls and Fear to Fall Assesment | Change from Baseline at 3 months, 6 months and 12 months.
  Questionnaire about, have fear to fall, since when, give up activities because of fear and since when. No puntuation.
Change Sun Expousure Questionnaire | Change from Baseline at 3 months, 6 months and 12 months.
  Questionnaire about hours expended outside, sun exposure and skin type. Only registration of data, without puntuations.
Change on Mediterranean Adherence Questionnaire PREDIMED | Change from Baseline at 3 months, 6 months and 12 months.
  14 items questionnaire about adherence to Mediterranean diet patron each question is puntuated with 1 (positive to mediterrranean diet) or 0. The total puntuation is a sum up from the 14 questions. Questions are about olive oil , vegetable and fruit , meat, desserts, wine, fish, and legumes consumption.
Changes on Mini Nutritional Assesment | Change from Baseline at 3 months, 6 months and 12 months.
  The MNA is a screening tool composed of two parts, 6 and 12 questions.First part permits detection of a decline in ingestion over the past three months (loss of appetite, decline of food intake, digestive problems, chewing or swallowing difficulties), weight loss in the past three months, current mobility impairment, an acute illness or major stress in the past three months, a neuropsychological problem (dementia or depression) and a decrease in body mass index (BMI). Second part of MNA evaluates living arrangements, the presence of polypharmacy or pressure ulcers, the number of full meals eaten daily, the amount and frequency of specific foods and fluids, and the mode of feeding. The patient reports nutritional and health status, and the practitioner determines weight and height (to calculate BMI), and mid-arm and mid-calf circumferences. The maximum score for first part is 14; a score of 12 points or greater means disorders.
Changes on ExernetElder questionnaire | Change from Baseline at 6 months and 12 months.
  Questionnaire about sociodemographic aspects such as participation on sports during lifespan, menarchy age and menopause age.
  Descriptive registration.
Change on Food Frequency Questionnaire | Baseline
  Food intake questionnaire (PREDIMED) asking about frequence of eating each food in last month. 139 different food from groups as daily products, eggs, meats and fishes, vegetables, fruits, legumes, fats and oils, desserts, miscalaneas and drinks. Each food could be answer with never, 1-3 a month, 1 a week, 2-4 a week, 5-6 a week, 1 a day, 2-3 a day, 4-6 a day, +6 a day.
  Each pint is registered but they do not pointed.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subias-Perie J, Navarrete-Villanueva D, Fernandez-Garcia AI, Moradell A, Alcala-Nalvaiz JT, Groessl EJ, Ara I, Vila-Maldonado S, Perez-Gomez J, Gonzalez-Gross M, Gomez-Cabello A, Vicente-Rodriguez G, Casajus JA. Cost-effectiveness of a multicomponent training programme for older adults with decreased functional capacity: An economic evaluation. Exp Gerontol. 2025 Nov;211:112911. doi: 10.1016/j.exger.2025.112911. Epub 2025 Sep 25. PMID 41015204
- [Derived] Moradell A, Iguacel I, Navarrete-Villanueva D, Fernandez-Garcia AI, Gonzalez-Gross M, Perez-Gomez J, Ara I, Casajus JA, Gomez-Cabello A, Vicente-Rodriguez G. Effects of a multicomponent training and a detraining period on cognitive and functional performance of older adults at risk of frailty. Aging Clin Exp Res. 2025 Apr 7;37(1):117. doi: 10.1007/s40520-025-03011-w. PMID 40192885
- [Derived] Subias-Perie J, Navarrete-Villanueva D, Fernandez-Garcia AI, Moradell A, Lozano-Berges G, Gesteiro E, Perez-Gomez J, Ara I, Gomez-Cabello A, Vicente-Rodriguez G, Casajus JA. Effects of a multicomponent training followed by a detraining period on metabolic syndrome profile of older adults. Exp Gerontol. 2024 Feb;186:112363. doi: 10.1016/j.exger.2024.112363. Epub 2024 Jan 19. PMID 38244708
- [Derived] Fernandez-Garcia AI, Moradell A, Navarrete-Villanueva D, Subias-Perie J, Perez-Gomez J, Ara I, Gonzalez-Gross M, Casajus JA, Vicente-Rodriguez G, Gomez-Cabello A. Effects of Multicomponent Training Followed by a Detraining Period on Frailty Level and Functional Capacity of Older Adults with or at Risk of Frailty: Results of 10-Month Quasi-Experimental Study. Int J Environ Res Public Health. 2022 Sep 29;19(19):12417. doi: 10.3390/ijerph191912417. PMID 36231712
- [Derived] Fernandez-Garcia AI, Gomez-Cabello A, Gomez-Bruton A, Moradell A, Navarrete-Villanueva D, Perez-Gomez J, Gonzalez-Gross M, Ara I, Casajus JA, Vicente-Rodriguez G. Effects of multicomponent training and detraining on the fitness of older adults with or at risk of frailty: results of a 10-month quasi-experimental study. Eur J Sport Sci. 2023 Aug;23(8):1696-1709. doi: 10.1080/17461391.2022.2104657. Epub 2022 Aug 11. PMID 35876120
- [Derived] Moradell A, Fernandez-Garcia AI, Navarrete-Villanueva D, Perez-Gomez J, Gesteiro E, Ara Royo I, Casajus JA, Gomez-Cabello A, Vicente-Rodriguez G. Does nutritional status influence the effects of a multicomponent exercise programme on body composition and physical fitness in older adults with limited physical function? Eur J Sport Sci. 2023 Jul;23(7):1375-1384. doi: 10.1080/17461391.2022.2092426. Epub 2022 Jul 11. PMID 35816744